CLINICAL TRIAL: NCT02655692
Title: CAP-Ketamine for Antidepressant Resistant PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); Brooke Army Medical Center (U.S. Federal Agency); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPLE-003-14W
Record Dates: First submitted 2016-01-07; First posted 2016-01-14 (Estimated); Results first posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: PTSD; Posttraumatic Stress Disorder
Keywords: PTSD; Ketamine; Veteran; Military; Clinical Trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Saline dose
  Interventions: Drug: Placebo/Saline
- Low Dose Ketamine (Experimental): Low Dose Ketamine (.20 mg/kg)
  Interventions: Drug: Ketamine
- High Dose Ketamine (Experimental): High Dose Ketamine (.50 mg/kg)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — FDA approved anesthetic medication with rapid acting antidepressant effects.
  Arms: High Dose Ketamine; Low Dose Ketamine
Drug: Placebo/Saline — This is a saline placebo/non-active solution.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety and efficacy of repeated doses of ketamine as compared to placebo, in reducing symptoms of Posttraumatic Stress Disorder (PTSD) in an active duty military and Veteran population.

DETAILED DESCRIPTION:
In this 2-site clinical trial, intended to evaluate the safety and efficacy of repeated doses of ketamine for treatment resistant PTSD, Veterans and active duty military personnel who meet criteria for PTSD and the additional inclusion and exclusion criteria will be randomized to one of three treatment arms (placebo, low dose ketamine, high dose ketamine). Participants receive the study drug via intravenous infusion twice per week for 4-weeks.

ELIGIBILITY:
Inclusion Criteria:

* male or female Veterans or active duty military personnel between the ages of 18 and 70 years
* diagnosis of PTSD
* history of trialing one or more antidepressant medications with little to no PTSD symptom improvement
* ability to provide written informed consent

Exclusion Criteria:

* females who are currently pregnant or breastfeeding
* current high risk for suicide
* history of severe head injury

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H. Krystal, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (3):
- United States (3):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Brooke Army Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdallah CG, Roache JD, Averill LA, Young-McCaughan S, Martini B, Gueorguieva R, Amoroso T, Southwick SM, Guthmiller K, Lopez-Roca AL, Lautenschlager K, Mintz J, Litz BT, Williamson DE, Keane TM, Peterson AL, Krystal JH; Consortium to Alleviate PTSD. Repeated ketamine infusions for antidepressant-resistant PTSD: Methods of a multicenter, randomized, placebo-controlled clinical trial. Contemp Clin Trials. 2019 Jun;81:11-18. doi: 10.1016/j.cct.2019.04.009. Epub 2019 Apr 15. PMID 30999057
- [Background] Abdallah CG, Roache JD, Gueorguieva R, Averill LA, Young-McCaughan S, Shiroma PR, Purohit P, Brundige A, Murff W, Ahn KH, Sherif MA, Baltutis EJ, Ranganathan M, D'Souza D, Martini B, Southwick SM, Petrakis IL, Burson RR, Guthmiller KB, Lopez-Roca AL, Lautenschlager KA, McCallin JP 3rd, Hoch MB, Timchenko A, Souza SE, Bryant CE, Mintz J, Litz BT, Williamson DE, Keane TM, Peterson AL, Krystal JH. Dose-related effects of ketamine for antidepressant-resistant symptoms of posttraumatic stress disorder in veterans and active duty military: a double-blind, randomized, placebo-controlled multi-center clinical trial. Neuropsychopharmacology. 2022 Jul;47(8):1574-1581. doi: 10.1038/s41386-022-01266-9. Epub 2022 Jan 19. PMID 35046508

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Saline dose
  Placebo: This is a saline placebo/non-active solution.
Period: Overall Study
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Started | 55 | 55 | 53
Completed | 36 | 41 | 40
Not Completed | 19 | 14 | 13

BASELINE CHARACTERISTICS:
Population: All available data was utilized in the analysis using raw means and SDs
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine | Total
Number analyzed (Participants) | 54 | 53 | 51 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (1.5) | 45 (1.5) | 43 (1.8) | 43.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 13 | 37
  Male | 40 | 43 | 38 | 121
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - non Hispanic | 37 | 28 | 29 | 94
  Black | 6 | 7 | 7 | 20
  Hispanic | 8 | 11 | 12 | 31
  Other | 3 | 7 | 3 | 13
PCL [Mean (Standard Deviation); unit: units on a scale] — The PTSD Checklist (PCL) is a brief measure of the symptoms of Posttraumatic Stress Disorder to measure change in PTSD symptoms. The PCL-5 is a 20-item self-report measure. A total symptom severity score (range - 0-80) with higher scores indicating greater severity.
  units on a scale | 51.95 (10.82) | 51.75 (12.38) | 50.23 (14.69) | 51.33 (12.62)

OUTCOME MEASURES:

1. Primary Outcome: PTSD Checklist (PCL)
Description: The PTSD Checklist (PCL) is a brief measure of the symptoms of Posttraumatic Stress Disorder (PTSD) to measure change in PTSD symptoms. The PCL-5 is a 20-item self-report measure, a total symptom severity score (range - 0-80) is obtained by summing the scores for each of the 20 items. (5-point Likert (0 = "Not at all" to 4 = "Extremely"). A total symptom severity score (range 0-80) with higher scores indicating greater severity for PTSD
Time Frame: Session 1 -Day 0
Population: The variability in the number of participants for data points resulted from a variety of reasons for example participants not showing up for appointments, dropping out of the study and/or illness.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 54 | 53 | 51
units on a scale | 48.56 (12.76) | 46.62 (17.71) | 47.88 (14.46)

2. Primary Outcome: The PTSD Checklist (PCL)
Description: as for outcome 1
Time Frame: Session 2 - Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 52 | 51 | 49
units on a scale | 37.65 (18.40) | 32.75 (19.39) | 30.10 (20.25)

3. Primary Outcome: The PTSD Checklist (PCL)
Description: as for outcome 1
Time Frame: Session 3 - Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 51 | 50 | 44
units on a scale | 36.90 (18.11) | 33.66 (18.67) | 34.20 (18.37)

4. Primary Outcome: The PTSD Checklist (PCL)
Description: as for outcome 1
Time Frame: Session 4 - Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 48 | 47 | 43
units on a scale | 34.75 (18.96) | 29.09 (20.61) | 32.58 (19.12)

5. Primary Outcome: The PTSD Checklist (PCL)
Description: as for outcome 1
Time Frame: Session 5 - Day 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 47 | 45 | 46
units on a scale | 35.11 (18.84) | 28.51 (21.12) | 31.46 (18.60)

6. Primary Outcome: The PTSD Checklist (PCL)
Description: as for outcome 1
Time Frame: Session 6 - Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 44 | 48 | 43
units on a scale | 30.80 (19.85) | 26.40 (21.12) | 27.91 (17.04)

7. Primary Outcome: The PTSD Checklist (PCL)
Description: as for outcome 1
Time Frame: Session 7 - Day 17
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 44 | 47 | 41
units on a scale | 28.48 (19.47) | 24.13 (20.15) | 26.54 (17.58)

8. Primary Outcome: The PTSD Checklist (PCL)
Description: as for outcome 1
Time Frame: Session 8 - Day 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 42 | 42 | 40
units on a scale | 29.31 (20.39) | 24.52 (20.45) | 26.73 (17.20)

9. Primary Outcome: The PTSD Checklist (PCL)
Description: as for outcome 1
Time Frame: Session 9 - Day 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 45 | 46 | 42
units on a scale | 28.31 (19.89) | 21.94 (20.35) | 25.62 (19.86)

10. Primary Outcome: The PTSD Checklist (PCL)
Description: as for outcome 1
Time Frame: Follow-up 1 - Day 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 44 | 43 | 41
units on a scale | 27.34 (20.25) | 21.35 (20.70) | 22.54 (17.98)

11. Primary Outcome: The PTSD Checklist (PCL)
Description: as for outcome 1
Time Frame: Follow-up 2 - Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 25 | 17 | 12
units on a scale | 37.84 (18.37) | 34.59 (18.45) | 39.58 (15.55)

12. Primary Outcome: The PTSD Checklist (PCL)
Description: as for outcome 1
Time Frame: Follow-up 3 - Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 24 | 18 | 11
units on a scale | 33.79 (19.80) | 33.72 (20.17) | 40.27 (16.29)

13. Primary Outcome: The PTSD Checklist (PCL)
Description: as for outcome 1
Time Frame: Follow-up 4 - Day 35
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 38 | 38 | 33
units on a scale | 26.92 (19.17) | 22.84 (21.46) | 24.09 (17.05)

14. Primary Outcome: The PTSD Checklist (PCL)
Description: as for outcome 1
Time Frame: Follow-up 5 - Day 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 35 | 39 | 37
units on a scale | 28.14 (20.92) | 25.62 (21.81) | 29.16 (19.85)

15. Primary Outcome: The PTSD Checklist (PCL)
Description: as for outcome 1
Time Frame: Follow-up 6 - Day 49
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 35 | 39 | 38
units on a scale | 30.71 (21.33) | 24.90 (20.66) | 30.21 (18.82)

16. Primary Outcome: The PTSD Checklist (PCL)
Description: as for outcome 1
Time Frame: Follow-up 7 - Day 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 39 | 41 | 35
units on a scale | 31.90 (21.08) | 24.32 (21.15) | 31.23 (19.81)

17. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Montgomery-Asberg Depression Rating Scale (MADRS) is a clinician rated ten-item diagnostic questionnaire to measure the severity of depression. The overall score ranges from 0 to 60 (0 to 6 - normal/symptom absent; 7 to 19 mild depression; 20 to 34 - moderate depression; >34 - severe depression)
Time Frame: Session 1 - Day 0
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 54 | 52 | 51
score on a scale | 28.24 (8.43) | 27.81 (10.30) | 27.84 (9.30)

18. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 17
Time Frame: Session 2 - Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 52 | 51 | 48
score on a scale | 17.75 (11.16) | 17.02 (13.02) | 12.94 (9.50)

19. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 17
Time Frame: Session 3 - Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 51 | 50 | 44
score on a scale | 19.98 (11.22) | 19.34 (12.77) | 17.86 (11.55)

20. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 17
Time Frame: Session 4 - Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 47 | 46 | 43
score on a scale | 19.94 (11.64) | 17.83 (13.11) | 18.54 (10.62)

21. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 17
Time Frame: Session 5 - Day 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 47 | 45 | 46
score on a scale | 20.70 (11.79) | 16.64 (12.90) | 18.07 (9.98)

22. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 17
Time Frame: Session 6 - Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 44 | 48 | 42
score on a scale | 18.36 (11.90) | 16.71 (13.47) | 16.83 (9.91)

23. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 17
Time Frame: Session 7 - Day 17
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 44 | 47 | 41
score on a scale | 17.02 (12.52) | 14.75 (12.98) | 15.15 (10.35)

24. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 17
Time Frame: Session 8 - Day 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 42 | 42 | 40
score on a scale | 17.02 (12.52) | 16.44 (13.66) | 15.78 (11.59)

25. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 17
Time Frame: Session 9 - Day 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 45 | 45 | 42
score on a scale | 17.11 (11.75) | 14.43 (12.29) | 14.24 (10.59)

26. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 17
Time Frame: Follow-up 1 - Day 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 44 | 42 | 41
score on a scale | 15.98 (12.32) | 12.91 (12.60) | 10.78 (9.85)

27. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 17
Time Frame: Follow-up 2 - Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 25 | 18 | 12
score on a scale | 24.00 (10.30) | 25.11 (12.20) | 25.08 (7.34)

28. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 17
Time Frame: Follow-up 3 - Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 24 | 17 | 11
score on a scale | 15.00 (11.55) | 19.18 (13.99) | 20.27 (8.32)

29. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 17
Time Frame: Follow-up 4 - Day 35
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 37 | 37 | 33
score on a scale | 16.08 (11.15) | 14.43 (12.71) | 12.72 (9.24)

30. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 17
Time Frame: Follow-up 5 - Day 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 35 | 39 | 36
score on a scale | 16.89 (12.51) | 15.74 (13.03) | 16.42 (9.39)

31. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 17
Time Frame: Follow-up 6 - Day 49
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 35 | 38 | 37
score on a scale | 19.60 (11.52) | 15.87 (11.79) | 17.68 (8.86)

32. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 17
Time Frame: Follow-up 7 - Day 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
Number analyzed (Participants) | 40 | 41 | 33
score on a scale | 19.45 (11.19) | 15.44 (12.98) | 19.58 (10.94)

ADVERSE EVENTS:
Time Frame: The study duration was 5 years; time Veterans participated was ~2 months total.
Arm/Group | Placebo | Low Dose Ketamine | High Dose Ketamine
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 0/53
Other Adverse Events (participants affected / at risk) | 25/55 | 42/55 | 38/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=55) | Low Dose Ketamine (N=55) | High Dose Ketamine (N=53)
agitation (Social circumstances) | 0 | 3 | 3
anxiety (Psychiatric disorders) | 0 | 2 | 2
diarrhea (Gastrointestinal disorders) | 2 | 3 | 2
fatigue (General disorders) | 2 | 3 | 4
headache (General disorders) | 7 | 14 | 6
irritability (Social circumstances) | 0 | 5 | 3
nausea/GI disturb (Gastrointestinal disorders) | 8 | 8 | 8
nightmares (General disorders) | 2 | 1 | 2
soreness/bruising at INJ site (General disorders) | 2 | 0 | 1
depression (Psychiatric disorders) | 1 | 1 | 1
suicidality (Psychiatric disorders) | 1 | 1 | 1
constipation (Gastrointestinal disorders) | 0 | 0 | 3
sweating (General disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT02655692/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT02655692/SAP_001.pdf